CLINICAL TRIAL: NCT02641457
Title: Intravitreal Aflibercept or Ranibizumab for Rubeosis Iridis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Olhos de Goiania (Other)
Responsible Party: Principal Investigator, Joao Nassaralla, Chairman, Instituto de Olhos de Goiania
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JN-015-2015
Record Dates: First submitted 2015-11-26; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Glaucoma; Rubeosis Iridis
Keywords: rubeosis iridis; glaucoma; ranibizumab; aflibercept
MeSH Terms: conditions — Glaucoma | interventions — aflibercept; Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aflibercept x Ranibizumab (Experimental): 12 eyes received an intraocular injection of 2.00 mg of aflibercept (IA) and 12 eyes patients received an intraocular injection of 1.25mg ranibizumab
  Interventions: Drug: Aflibercept; Drug: Ranibizumab

INTERVENTIONS:
Drug: Aflibercept — 12 eyes received an intraocular injection of 2.00 mg of aflibercept (IA) and IOP were measured by tonometer. The neovascularization was evaluated by biomicroscope.
  Other Names: Eylea
Drug: Ranibizumab — 12 eyes received an intraocular injection of 1.25mg ranibizumab and IOP were measured by tonometer. The neovascularization was evaluated by biomicroscope.
  Other Names: Lucentis

SUMMARY:
Aflibercept (Eylea®) and ranibizumab (Lucentis®) are an anti-VEGF, but there are differences between the two drugs. To determine and compare whether intraocular aflibercept and ranibizumab decreases rubeosis iridis (RI) in patients with neovascular glaucoma (NVG).

DETAILED DESCRIPTION:
Aflibercept (Eylea®) and ranibizumab (Lucentis®) are an anti-VEGF, but there are differences between the two drugs. Lucentis is administered in the form of smaller molecules, which is thought to give Lucentis an advantage over Eylea in its ability to penetrate the eye's retina and halt abnormal blood vessel growth contributing to advanced macular degeneration and scarring that causes blindness. They may have a role in treating ocular disorders involving fibrovascular proliferation. To determine and compare whether intraocular aflibercept and ranibizumab decreases rubeosis iridis (RI) in patients with neovascular glaucoma (NVG).

ELIGIBILITY:
Criteria:

Inclusion Criteria:

* Ability to provide written informed consent and comply with study assessments for the full duration of the study
* Age > 18 years
* Ischemic central retina vein occlusion (CRVO) within 3 months of enrollment as per the following inclusion criteria
* Three of the following clinical tests must be present to demonstrate ischemic CRVO
* Visual Acuity 20/200 or worse
* Loss of 1-2e isopter on Goldmann Visual field (Kwon et al. 2001)
* Electroretinogram demonstrating b wave amplitude less than 60% of A wave.

Exclusion Criteria:

* Angle neovascularization greater than 3 clock hours with IOP over 30 (Neovascular glaucoma)
* Any previous retinal laser photocoagulation to the study eye
* Any previous intravitreal injection in study eye (triamcinolone or other)
* Any previous vitrectomy in study eye (posterior or anterior associated with vitreous loss in cataract surgery)
* Intracapsular cataract extraction (posterior capsule needs to be present)
* Previous history of retinal detachment in study eye
* Any previous radiation treatments to head/ neck
* Inability to assess iris neovascularization (corneal opacity precluding gonioscopy)
* Significant cardiovascular disease or cancer that would prevent follow-up visits or completion of the 12 month study
* Significant diabetic retinopathy in the fellow eye (diabetic macular edema, proliferative diabetic retinopathy, or high-risk non-proliferative diabetic retinopathy)
* Pregnancy (positive pregnancy test)
* Prior enrollment in any study for vein occlusion in the study eye
* Participation in another simultaneous medical investigator or trial Ocular disorders in the study eye that may confound interpretation of study results, including retinal detachment, macular hole, or choroidal neovascularization of any cause (e.g., DME AMD, ocular histoplasmosis, or pathologic myopia)
* Concurrent disease in the study eye that could compromise visual acuity or require medical or surgical intervention during the study period
* Aphakia or absence of the posterior capsule in the study eye
* Previous violation of the posterior capsule is also excluded unless it occurred as a result of YAG laser posterior capsulotomy in association with prior, posterior chamber intraocular lens implantation
* History of idiopathic or autoimmune uveitis in either eye Structural damage to the center of the macula in the study eye preexisting to CRVO likely to preclude improvement in visual acuity following the resolution of macular edema, including atrophy of the retinal pigment epithelium, subretinal fibrosis, laser scar(s)
* Vitreomacular traction or epiretinal membrane in the study eye evident biomicroscopically or by OCT
* Ocular inflammation (including trace or above) in the study eye Uncontrolled glaucoma (defined as intraocular pressure ≥30 mm Hg despite treatment with anti- medications) or previous filtration surgery in the study eye Systemic Conditions
* Uncontrolled Blood pressure exceeding diastolic pressure of 100 mm Hg (sitting) during the screening period
* Uncontrolled diabetes mellitus
* Renal failure requiring dialysis or renal transplant
* Premenopausal women not using adequate contraception
* Previous participation in other studies of investigational drugs (excluding vitamins and minerals) within 3 months preceding Day 0
* History of other disease, metabolic dysfunction, physical examination finding, or other findings giving reasonable suspicion of a disease or condition that contraindicates the use an investigational drug, might affect interpretation of the results of the study, or render the subject at high risk from treatment complications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Degree of rubeosis iridis by biomicroscope | 1 year follow up
  Compare results of rubeosis iridis regression after aflibercept or ranibizumab intraocular injection with decrease neovascularization - 1 year follow up
Degree of rubeosis iridis assessed by intraocular pressure | 1 year follow up
  Compare results of rubeosis iridis regression after aflibercept or ranibizumab intraocular injection with decrease intraocular pressure (IOP) - 1 year follow up

CONTACTS AND LOCATIONS:
Overall Officials: Joao J Nassaralla, MD PhD, Study Chair — Instituto de Olhos de Goiânia
Locations (1):
- Instituto de Olhos de Goiania, Goiânia, Goiás, Brazil